CLINICAL TRIAL: NCT00597012
Title: Partial Meniscectomy Versus Nonoperative Management in Meniscal Tear With OA: A Randomized Controlled Trial (MeTeOR)
Brief Title: Comparing Surgery Versus Standard Physical Therapy in Treating People With a Meniscal Tear and Osteoarthritis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Jeffrey Neil Katz, MD, Professor of Medicine and Orthopedic Surgery, Harvard Medical School; Director, Orthopaedic and Arthritis Center for Outcomes Research, Brigham & Women's Hospital, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01AR055557 (NIH)
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Results first posted 2014-01-27 (Estimated); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Osteoarthritis
Keywords: Meniscal Tear; Osteoarthritis; Arthroscopic Partial Meniscectomy; Physical Therapy; Total Knee Arthroplasty; Total Knee Replacement
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgical (Experimental): Participants will undergo arthroscopic partial menisectomy (APM) surgery and offered postoperative rehabilitative physical therapy.
  Interventions: Procedure: Arthroscopic partial menisectomy; Other: Postoperative rehabilitative physical therapy
- Nonoperative (Active Comparator): Participants will undergo standard physical therapy that will include strengthening and stretching sessions one to three times a week for 8 weeks.
  Interventions: Other: Standard physical therapy

INTERVENTIONS:
Procedure: Arthroscopic partial menisectomy — Arthroscopic partial meniscectomy is a surgical procedure that is performed to remove a piece of torn cartilage in the knee joint. Incisions for arthroscopy are quite small, usually about 1 centimeter each. The torn meniscus can be removed using a number of different instruments, including small shavers and scissors.
  Arms: Surgical
Other: Standard physical therapy — Participants will undergo standard physical therapy that will include strengthening and stretching sessions one to three times a week for 8 weeks. This physical therapy regimen will have similar elements and goals as the postoperative intervention offered to Group 1 participants.
  Arms: Nonoperative
Other: Postoperative rehabilitative physical therapy — This physical therapy is geared specifically toward rehabilitation after APM surgery.
  Arms: Surgical

SUMMARY:
There are two cartilage structures, called menisci, in each knee joint. A torn meniscus can be caused by a traumatic injury or aging-related degeneration. Osteoarthritis (OA) is a type of arthritis that is caused by the breakdown and eventual loss of another type of cartilage that covers the end of bones within a joint. In people who have knee OA, a meniscal tear can easily lead to disability. This study will compare the effectiveness of two recommended treatments, surgery and physical therapy, for people with a torn meniscus and knee OA.

DETAILED DESCRIPTION:
OA is the most common form of arthritis in the United States. Symptoms of knee OA include pain in and around the knee that typically worsens with weight-bearing activities, morning stiffness, and tenderness. A person with OA who experiences a torn meniscus--a cartilage structure within the knee that provides stability and proper weight distribution--is especially at risk for disability. Past studies have shown that arthroscopic partial meniscectomy (APM), a type of knee surgery, usually relieves symptoms and improves function in people suffering from a meniscal tear. However, the success of APM is more variable among people with already existing OA. Clinicians are also uncertain about the short- and long-term benefits, drawbacks, and indications for APM in people with OA and meniscal tears. The purpose of this study is to compare the effectiveness of two treatments, APM surgery and standard physical therapy, for people with OA and a torn meniscus.

This study will last 12 years. At the initial study visit, participants will be randomly assigned to one of two groups.

* Group 1 participants will undergo APM surgery at a time that is convenient for the participant and surgeon. After surgery, participants will be referred for rehabilitative physical therapy to regain strength and flexibility of the knee. For participants who choose to do physical therapy, the duration of treatment will depend on individual progress.
* Group 2 participants will receive standard physical therapy to increase strength and flexibility of the knee. This will include one to three weekly exercise sessions over an 8-week period.

The study consists of up to 5 visits to the center:

* Visit 1, the enrollment visit: sign the consent form, fill out a questionnaire, have a physical examination of the knee and find out your treatment group (surgery or physical therapy
* Visit 2, at 3 months after enrollment: Fill out a questionnaire and have a physical examination of the knee
* Visit 3, at 18 months: Fill out a questionnaire, have an MRI of the knee (if eligible) and xrays of both knees
* Visit 4, at 5 years: Fill out a questionnaire, have an MRI of the knee (if eligible) and xrays of both knees
* Visit 5, at 12 years: Fill out a questionnaire, have a physical examination of the knee, have an MRI of the knee (if eligible) and xrays of both knees

Telephone calls: During the first 3 months of the study, all participants will receive check-up phone calls every 2 weeks, followed by quarterly phone calls for the initial 2 years in the study

Questionnaires: Participants will also complete mailed questionnaires at 6 months, and 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, and 12 years after enrollment. The questionnaires will include questions about knee pain, ability to walk, recreational activities, general health, and satisfaction with with treatment.

ELIGIBILITY:
Inclusion Criteria:

* OA symptoms lasting at least 1 month and managed with medications, activity limitations, and/or physical therapy
* At least one symptom consistent with a torn meniscus. Symptoms may include clicking, catching, popping, giving way, pain with pivot or torque, episodic pain, and/or pain that is acute and localized to one joint line.
* Available knee X-ray (within 6 months) and MRI (within 3 years)
* Evidence of osteophyte formation or cartilage fissure, tear, or loss on a knee MRI OR plain radiographic evidence of osteophyte formation or joint space narrowing
* Evidence of a meniscal tear (tear extending to surface of meniscus) on a knee MRI
* Willingness to undergo random assignment and sign an informed consent

Exclusion Criteria:

* Chronically locked knee
* Kellgren-Lawrence Grade IV status, indicating advanced OA and usually the need for total knee replacement
* Contraindication to MRI
* Radiographic chondrocalcinosis (a condition in which there are deposits of calcium pyrophosphate dihydrate [CPPD] crystals in one or more joints that eventually result in damage to the affected joints) AND acute symptomatic pseudogout
* Inflammatory diseases (e.g., rheumatoid arthritis, psoriatic arthritis, systemic lupus erythematosus, gout, pseudogout)
* Injection with viscosupplementation in the affected knee in the 4 weeks before study entry
* Any medical contraindications to surgery or physical therapy
* Both knees are symptomatic for meniscal tears and a candidate for bilateral APMs
* Prior surgery on an affected knee
* Pregnancy or possible pregnancy
* Claim filed for worker's compensation
* Unable or unwilling to give informed consent
* Unable or unwilling to attend physical therapy sessions at designated locations or in the community

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2008-05; Primary Completion 2012-02 (Actual); Study Completion 2025-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey N. Katz, MD, MS, Principal Investigator — Brigham and Women's Hospital
Locations (7):
- United States (7):
  - Rush University Medical Center, Chicago, Illinois
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University in St Louis, School of Medicine, St Louis, Missouri
  - Hospital for Special Surgery, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Katz JN, Chaisson CE, Cole B, Guermazi A, Hunter DJ, Jones M, Levy BA, Mandl LA, Martin S, Marx RG, Safran-Norton C, Roemer FW, Skoniecki D, Solomon DH, Spindler KP, Wright J, Wright RW, Losina E. The MeTeOR trial (Meniscal Tear in Osteoarthritis Research): rationale and design features. Contemp Clin Trials. 2012 Nov;33(6):1189-96. doi: 10.1016/j.cct.2012.08.010. Epub 2012 Sep 5. PMID 22968127
- [Background] Katz JN, Brophy RH, Chaisson CE, de Chaves L, Cole BJ, Dahm DL, Donnell-Fink LA, Guermazi A, Haas AK, Jones MH, Levy BA, Mandl LA, Martin SD, Marx RG, Miniaci A, Matava MJ, Palmisano J, Reinke EK, Richardson BE, Rome BN, Safran-Norton CE, Skoniecki DJ, Solomon DH, Smith MV, Spindler KP, Stuart MJ, Wright J, Wright RW, Losina E. Surgery versus physical therapy for a meniscal tear and osteoarthritis. N Engl J Med. 2013 May 2;368(18):1675-84. doi: 10.1056/NEJMoa1301408. Epub 2013 Mar 18. PMID 23506518
- [Background] Deshpande BR, Losina E, Smith SR, Martin SD, Wright RJ, Katz JN. Association of MRI findings and expert diagnosis of symptomatic meniscal tear among middle-aged and older adults with knee pain. BMC Musculoskelet Disord. 2016 Apr 11;17:154. doi: 10.1186/s12891-016-1010-2. PMID 27067990
- [Background] Tuakli-Wosornu YA, Selzer F, Losina E, Katz JN. Predictors of Exercise Adherence in Patients With Meniscal Tear and Osteoarthritis. Arch Phys Med Rehabil. 2016 Nov;97(11):1945-1952. doi: 10.1016/j.apmr.2016.05.011. Epub 2016 Jun 11. PMID 27296899
- [Background] Katz JN, Wright J, Spindler KP, Mandl LA, Safran-Norton CE, Reinke EK, Levy BA, Wright RW, Jones MH, Martin SD, Marx RG, Losina E. Predictors and Outcomes of Crossover to Surgery from Physical Therapy for Meniscal Tear and Osteoarthritis: A Randomized Trial Comparing Physical Therapy and Surgery. J Bone Joint Surg Am. 2016 Nov 16;98(22):1890-1896. doi: 10.2106/JBJS.15.01466. PMID 27852905
- [Background] Katz JN, Smith SR, Yang HY, Martin SD, Wright J, Donnell-Fink LA, Losina E. Value of History, Physical Examination, and Radiographic Findings in the Diagnosis of Symptomatic Meniscal Tear Among Middle-Aged Subjects With Knee Pain. Arthritis Care Res (Hoboken). 2017 Apr;69(4):484-490. doi: 10.1002/acr.22975. Epub 2017 Mar 3. PMID 27390312
- [Background] MacFarlane LA, Yang H, Collins JE, Guermazi A, Jones MH, Teeple E, Xu L, Losina E, Katz JN. Associations among meniscal damage, meniscal symptoms and knee pain severity. Osteoarthritis Cartilage. 2017 Jun;25(6):850-857. doi: 10.1016/j.joca.2016.12.023. Epub 2016 Dec 30. PMID 28043939
- [Background] Winter AR, Collins JE, Katz JN. The likelihood of total knee arthroplasty following arthroscopic surgery for osteoarthritis: a systematic review. BMC Musculoskelet Disord. 2017 Oct 4;18(1):408. doi: 10.1186/s12891-017-1765-0. PMID 28978308
- [Background] Luc-Harkey BA, Safran-Norton CE, Mandl LA, Katz JN, Losina E. Associations among knee muscle strength, structural damage, and pain and mobility in individuals with osteoarthritis and symptomatic meniscal tear. BMC Musculoskelet Disord. 2018 Jul 27;19(1):258. doi: 10.1186/s12891-018-2182-8. PMID 30049269
- [Background] MacFarlane LA, Yang H, Collins JE, Jarraya M, Guermazi A, Mandl LA, Martin SD, Wright J, Losina E, Katz JN; MeTeOR Investigator Group. Association of Changes in Effusion-Synovitis With Progression of Cartilage Damage Over Eighteen Months in Patients With Osteoarthritis and Meniscal Tear. Arthritis Rheumatol. 2019 Jan;71(1):73-81. doi: 10.1002/art.40660. Epub 2018 Nov 29. PMID 30133187
- [Background] MacFarlane LA, Yang H, Collins JE, Guermazi A, Jones MH, Spindler KP, Winter AR, Losina E, Katz JN; the MeTeOR Investigator Group; Brophy RH, Cole BJ, Levy BA, Mandl LA, Martin S, Marx RG, Matava M, Safran-Norton C, Stuart M, Wright R. Influence of Baseline Magnetic Resonance Imaging Features on Outcome of Arthroscopic Meniscectomy and Physical Therapy Treatment of Meniscal Tears in Osteoarthritis. Am J Sports Med. 2019 Mar;47(3):612-619. doi: 10.1177/0363546518819444. Epub 2019 Jan 17. PMID 30653921
- [Background] MacFarlane LA, Yang H, Collins JE, Guermazi A, Mandl LA, Levy BA, Marx RG, Safran-Norton CE, Losina E, Katz JN; Meniscal Tear in Osteoarthritis Research Investigator Group. Relationship Between Patient-Reported Swelling and Magnetic Resonance Imaging-Defined Effusion-Synovitis in Patients With Meniscus Tears and Knee Osteoarthritis. Arthritis Care Res (Hoboken). 2019 Mar;71(3):385-389. doi: 10.1002/acr.23592. PMID 29726627
- [Background] Collins JE, Losina E, Marx RG, Guermazi A, Jarraya M, Jones MH, Levy BA, Mandl LA, Martin SD, Wright RW, Spindler KP, Katz JN; MeTeOR Investigator Group. Early Magnetic Resonance Imaging-Based Changes in Patients With Meniscal Tear and Osteoarthritis: Eighteen-Month Data From a Randomized Controlled Trial of Arthroscopic Partial Meniscectomy Versus Physical Therapy. Arthritis Care Res (Hoboken). 2020 May;72(5):630-640. doi: 10.1002/acr.23891. PMID 30932360
- [Background] Katz JN, Shrestha S, Losina E, Jones MH, Marx RG, Mandl LA, Levy BA, MacFarlane LA, Spindler KP, Silva GS; METEOR Investigators; Collins JE. Five-Year Outcome of Operative and Nonoperative Management of Meniscal Tear in Persons Older Than Forty-Five Years. Arthritis Rheumatol. 2020 Feb;72(2):273-281. doi: 10.1002/art.41082. Epub 2019 Dec 15. PMID 31429198
- [Derived] Collins JE, Shrestha S, Losina E, Marx RG, Guermazi A, Jarraya M, Jones MH, Levy BA, Mandl LA, Williams EE, Wright RW, Spindler KP, Katz JN; METEOR Investigator Group. Five-Year Structural Changes in the Knee Among Patients With Meniscal Tear and Osteoarthritis: Data From a Randomized Controlled Trial of Arthroscopic Partial Meniscectomy Versus Physical Therapy. Arthritis Rheumatol. 2022 Aug;74(8):1333-1342. doi: 10.1002/art.42105. Epub 2022 Jun 28. PMID 35245416
- [Derived] Katz JN, Collins JE, Jones M, Spindler KP, Marx RG, Mandl LA, Levy BA, Wright R, Jarraya M, Guermazi A, MacFarlane LA, Losina E, Chang Y. Association Between Structural Change Over Eighteen Months and Subsequent Symptom Change in Middle-Aged Patients Treated for Meniscal Tear. Arthritis Care Res (Hoboken). 2023 Feb;75(2):340-347. doi: 10.1002/acr.24796. Epub 2022 Oct 21. PMID 34606692
- [Derived] MacFarlane LA, Yang H, Collins JE, Brophy RH, Cole BJ, Spindler KP, Guermazi A, Jones MH, Mandl LA, Martin S, Marx RG, Levy BA, Stuart M, Safran-Norton C, Wright J, Wright RW, Losina E, Katz JN. Association Between Baseline Meniscal Symptoms and Outcomes of Operative and Nonoperative Treatment of Meniscal Tear in Patients With Osteoarthritis. Arthritis Care Res (Hoboken). 2022 Aug;74(8):1384-1390. doi: 10.1002/acr.24588. Epub 2022 May 6. PMID 33650303

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Meniscal Tear in Osteoarthritis Research (MeTeOR) trial was performed in seven academic referral centers with enrollment occurring from June 2008 through August 2011.
Groups:
- Arthroscopic Partial Meniscectomy (APM): Participants underwent arthroscopic partial menisectomy (APM) surgery and were offered postoperative rehabilitative physical therapy.
- Physical Therapy (PT): Participants underwent standard physical therapy that included strengthening and stretching sessions one to three times a week for 8 weeks.
Period: Overall Study
Arm/Group | Arthroscopic Partial Meniscectomy (APM) | Physical Therapy (PT)
Started | 174 | 177
Completed | 161 | 169
Not Completed | 13 | 8
Not completed — Death | 1 | 1
Not completed — Underwent Total Knee Replacement (TKR) | 3 | 1
Not completed — Withdrawal by Subject | 7 | 4
Not completed — Ineligible | 2 | 0
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Population: Analysis was completed on the 330 active participants in the study at 6 months.
Groups:
- Arthroscopic Partial Meniscectomy: Participants will undergo arthroscopic partial menisectomy (APM) surgery and offered postoperative rehabilitative physical therapy.
- Physical Therapy: Participants will undergo standard physical therapy that will include strengthening and stretching sessions one to three times a week for 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Arthroscopic Partial Meniscectomy | Physical Therapy | Total
Number analyzed (Participants) | 161 | 169 | 330
Age, Customized [Mean (Standard Deviation); unit: years] | 59.0 (7.9) | 57.8 (6.8) | 58.4 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 97 | 187
  Male | 71 | 72 | 143
Race/Ethnicity, Customized [Number; unit: participants]
  White | 138 | 142 | 280
  Black or African American | 15 | 17 | 32
  Hispanic | 2 | 5 | 7
  Other | 6 | 5 | 11
Index Knee [Number; unit: participants]
  Right | 70 | 68 | 138
  Left | 91 | 101 | 192
Mean Body-Mass Index [Mean (Standard Deviation); unit: kg/m^2] — The body-mass index is the weight in kilograms divided by the square of the height in meters.
  kg/m^2 | 30.0 (6.1) | 30.0 (6.1) | 30.0 (6.1)
WOMAC physical-function score [Mean (Standard Deviation); unit: Units on a scale] — Scores on the physical-function subscale of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) range from 0 to 100, with higher scores indicating more limitation of physical function.
  Units on a scale | 37.1 (17.9) | 37.5 (18.3) | 37.3 (18.1)
KOOS pain score [Mean (Standard Deviation); unit: Units on a scale] — Scores on the pain scale of the Knee Injury and Osteoarthritis Outcome Scale (KOOS) range from 0 to 100, with higher scores indicating more pain.
  Units on a scale | 46.0 (15.5) | 47.2 (16.4) | 46.6 (16.0)
Mental Health Index 5 score [Mean (Standard Deviation); unit: Units on a scale] — Scores on the Mental Health Index 5 range from 0 to 100, with higher scores indicating better mental health.
  Units on a scale | 74.8 (12.9) | 74.0 (13.9) | 74.4 (13.5)
SF-36 Physical Activity score [Mean (Standard Deviation); unit: Units on a scale] — Scores on the physical-activity scale of the Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36) range from 0 to 100, with higher scores indicating greater physical activity.
  Units on a scale | 44.3 (23.7) | 43.3 (23.3) | 43.8 (23.5)
Kellgren-Lawrence grade [Number; unit: participants] — A Kellgren-Lawrence grade of 0 (no osteophytes or joint-space narrowing) indicates no osteoarthritis, a grade of 1 (questionable osteophyte) indicates possible osteoarthritis; a grade of 2 (definite osteophyte, no joint-space narrowing) indicates mild osteoarthritis, a grade of 3 (less than or equal to 50% joint-space narrowing) indicates moderate osteoarthritis, and a grade of 4 (greater than 50% joint-space narrowing) indicates severe osteoarthritis.
  Total number of participants analyzed does not equal the total number of participants due to missing data.
  participants
    0 | 34 | 36 | 70
    1 | 26 | 35 | 61
    2 | 37 | 39 | 76
    3 | 45 | 39 | 84

OUTCOME MEASURES:

1. Primary Outcome: WOMAC Functional Status - Difference From Baseline
Description: Scores on the physical-function subscale of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) range from 0 to 100, with higher scores indicating more limitation of physical function. The primary outcome was the difference between the study groups with respect to the change in the score on the physical-function scale of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) from baseline to 6 months after randomization.
Time Frame: Baseline and 6 months
Measure: Mean (95% Confidence Interval); unit: Score
Groups:
- Arthroscopic Partial Meniscectomy: Participants underwent arthroscopic partial menisectomy (APM) surgery and were referred for postoperative rehabilitative physical therapy.
- Physical Therapy: Participants underwent standard physical therapy that included strengthening and stretching sessions one to three times a week for 8 weeks.
Arm/Group | Arthroscopic Partial Meniscectomy | Physical Therapy
Number analyzed (Participants) | 161 | 169
Score | 20.9 [17.9 to 23.9] | 18.5 [15.6 to 21.5]
Statistical Analysis 1: Comparison: Arthroscopic Partial Meniscectomy vs Physical Therapy; The primary analysis was implemented with an analysis of covariance with changes in the WOMAC physical-function score from baseline to 6 months as the dependent variable, treatment as the independent variable of interest, and study site as a covariate. The primary analysis used a modified intention-to-treat approach in which patients who did not withdraw from the study were evaluated in the group to which they were randomly assigned; Test type: Superiority or Other; p = 0.26, ANCOVA; Mean Difference (Final Values) = 2.4, 95% CI 2-sided [-1.8 to 6.5]

2. Secondary Outcome: KOOS Pain - Difference From Baseline
Description: Scores on the pain scale of the Knee Injury and Osteoarthritis Outcome Scale (KOOS) range from 0 to 100, with higher scores indicating more pain. The secondary outcome was the difference between the study groups with respect to the change in the score on the pain scale of the Knee Injury and Osteoarthritis Outcome Scale (KOOS) from baseline to 6 months after randomization.
Time Frame: Baseline to 6 months
Measure: Mean (95% Confidence Interval); unit: Score
Arm/Group | Arthroscopic Partial Meniscectomy | Physical Therapy
Number analyzed (Participants) | 161 | 169
Score | 24.2 [21.3 to 27.1] | 21.3 [18.4 to 24.2]
Statistical Analysis 1: Comparison: Arthroscopic Partial Meniscectomy vs Physical Therapy; Test type: Superiority or Other; p = 0.16, ANCOVA; Mean Difference (Final Values) = 2.9, 95% CI 2-sided [-1.2 to 7.0]

3. Secondary Outcome: SF-36 Physical Functional Status Scale - Difference From Baseline
Description: Scores on the physical-activity scale of the Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36) range from 0 to 100, with higher scores indicating greater physical activity.
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: Score
Arm/Group | Arthroscopic Partial Meniscectomy | Physical Therapy
Number analyzed (Participants) | 161 | 169
Score | 24.2 [20.3 to 28.0] | 23.1 [19.2 to 27.0]
Statistical Analysis 1: Comparison: Arthroscopic Partial Meniscectomy vs Physical Therapy; Test type: Superiority or Other; p = 0.68, ANCOVA; Mean Difference (Net) = 1.1, 95% CI 2-sided [-4.4 to 6.6]

4. Secondary Outcome: Total Knee Replacement - Subjects Received
Description: Number of subjects that elected to undergo Total Knee Replacement or Total Knee Arthroplasty between baseline and 60 month follow up. Intended to show the total number of participants that underwent Total Knee Replacement in the period following the initial intervention through 60 month follow up.
Time Frame: Baseline to 60 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arthroscopic Partial Meniscectomy | Physical Therapy
Number analyzed (Participants) | 161 | 169
Participants | 16 | 9

5. Secondary Outcome: KOOS Pain - Mean at 60 Months
Description: Scores on the pain scale of the Knee Injury and Osteoarthritis Outcome Scale (KOOS) range from 0 to 100, with higher scores indicating more pain. The secondary outcome was the mean KOOS pain for each of the study groups 60 months after randomization.
Time Frame: 60 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arthroscopic Partial Meniscectomy (APM) | Physical Therapy (PT)
Number analyzed (Participants) | 161 | 169
score on a scale | 18.2 [15.4 to 20.9] | 19.4 [16.7 to 22.1]

ADVERSE EVENTS:
Time Frame: 60 months
Groups:
- Arthroscopic Partial Meniscectomy: Participants underwent arthroscopic partial menisectomy (APM) surgery and were offered postoperative rehabilitative physical therapy.
Arm/Group | Arthroscopic Partial Meniscectomy | Physical Therapy
All-Cause Mortality (participants affected / at risk) | 1/174 | 1/177
Serious Adverse Events (participants affected / at risk) | 3/174 | 2/177
Other Adverse Events (participants affected / at risk) | 15/174 | 13/177
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arthroscopic Partial Meniscectomy (N=174) | Physical Therapy (N=177)
Cardiovascular (Cardiac disorders) | 2 (2) | 2 (2)
Hypoxemia (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arthroscopic Partial Meniscectomy (N=174) | Physical Therapy (N=177)
Muskuloskeletal (Musculoskeletal and connective tissue disorders) | 7 (7) | 6 (6)
Pain in the back, hip, or foot (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Cardiovascular (Cardiac disorders) | 6 (6) | 3 (3)

LIMITATIONS AND CAVEATS:
Surgical randomized controlled trials present methodological challenges, including crossover from one group to the other.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No